CLINICAL TRIAL: NCT02883608
Title: Cap Assisted Forward-Viewing Endoscope vs Side-Viewing Endoscope for Examination of Major Duodenal Papilla
Acronym: KappaII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Mohamed Abdelhafez, Cap Assisted Forward-Viewing Endoscope vs Side-Viewing Endoscope for Examination of Major Duodenal Papilla, Technical University of Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 216/16 s
Record Dates: First submitted 2016-08-21; First posted 2016-08-30 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Duodenal Papilla, Major
Keywords: Papilla; major duodenal papilla; ampulla of vater

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial cap assisted endoscopy (Experimental): undergo initial cap assisted forward-viewing endoscope then side-viewing duodenoscope
  Interventions: Procedure: cap assisted forward-viewing endoscope
- Initial standard endoscopy (Active Comparator): undergo initial side-viewing duodenoscope then cap assisted forward-viewing endoscope
  Interventions: Procedure: cap assisted forward-viewing endoscope

INTERVENTIONS:
Procedure: cap assisted forward-viewing endoscope — a cap fitted to the to top of the forward-viewing endoscope

SUMMARY:
Examination of major duodenal papilla (MDP) using a standard forward-viewing esophagogastroduodenoscopy (S-EGD) is limited. Until now, side-viewing duodenoscope is the modality of choice to examine the MDP. Cap assisted esophagogastroduodenoscopy (CA-EGD) uses a cap fitted to the tip of the scope that can depress the mucosal folds and thus improve visualization and examination of MDP. The aim of this study is to compare CA-EGD to side*viewing duodenoscope for complete examination of MDP.

ELIGIBILITY:
Inclusion Criteria:

* indication for elective upper endoscopy
* age over 18 years
* ability to provide informed consent

Exclusion Criteria:

* surgically altered upper gastrointestinal tract
* known or suspected upper gastrointestinal strictures
* upper gastrointestinal bleeding
* biliary stent
* planned endoscopic intervention
* American Society of Anesthesiologists class III or higher
* contraindication for or refusal of sedation with Propofol
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2017-01-22 (Actual)

PRIMARY OUTCOMES:
Rate of complete visualisation of papilla duodeni major | within 5 minutes after intubation of the esophagus
  complete visualization is defined by visualization of both proximal and distal ends together with the orifice of the papilla

SECONDARY OUTCOMES:
Duration needed to localize the papilla | within 5 minutes after intubation of the esophagus

CONTACTS AND LOCATIONS:
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelhafez M, Phillip V, Hapfelmeier A, Sturm V, Elnegouly M, Dollhopf M, Kassem A, Klare P, Nennstiel S, Schmid RM, von Delius S, Eckel F. Comparison of cap-assisted endoscopy vs. side-viewing endoscopy for examination of the major duodenal papilla: a randomized, controlled, noninferiority crossover study. Endoscopy. 2019 May;51(5):419-426. doi: 10.1055/a-0662-5445. Epub 2018 Sep 10. PMID 30199900